CLINICAL TRIAL: NCT00492570
Title: GER-009-06-AVX Early Therapy in Multiple Sclerosis
Acronym: FIT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Other Study IDs: GER-009-06-AVX
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive Dysfunction in Multiple sclerosis; early treatment; Avonex; interferon beta 1a; Cognitive Dysfunction
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to increase awareness for early therapy with Avonex for Multiple Sclerosis (MS) and the cognitive dysfunction that accompanies MS, and to record safety data for Avonex.

DETAILED DESCRIPTION:
This study will address the cognitive dysfunction associated with MS. It will track these changes and show that early intervention with Avonex is effective in slowing MS and its effect on patients. Safety data will also be collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* CIS (according to indication) or early Relapsing Remitting Multiple Sclerosis

Exclusion Criteria:

* treatment with DMT during the last 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: multi-center using 150-200 neurologists and their patient populations.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Study Director, Principal Investigator — Biogen